CLINICAL TRIAL: NCT05132400
Title: The Implementation of Psychologically Informed Physical Therapy to Prevent Chronification in Service Members With Musculoskeletal Disorders
Brief Title: PiPT in ADSM With MSD
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); United States Naval Medical Center, Portsmouth (U.S. Federal Agency); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 21-01351
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain; Musculoskeletal Diseases or Conditions
Keywords: Psychologically informed Physical Therapy (PiPT)
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Training Arm (Control): To receive physical therapy treatment as usual, before PiPT occurs
- Post-Training Arm (Intervention)
  Interventions: Behavioral: Psychological-informed Physical Therapy (PiPT) Training

INTERVENTIONS:
Behavioral: Psychological-informed Physical Therapy (PiPT) Training — An approach designed to incorporate the concepts of cognitive behavioral therapy (CBT) for pain management into routine clinical PT practice in order to modify maladaptive responses associated with chronicity. The goal of PiPT is to promote a fast and optimal recovery by removing psychological obstacles, obviating the need for referral to a psychologist and facilitating triage to other health professionals in a timely manner when needed. PiPT training includes education about the neuropsychology of pain, patient communication skills, and identification of psychosocial risk factors for chronicity and treatment approaches that include reassurance, relaxation, and psycho-behavioral reactivation.
  Groups: Post-Training Arm (Intervention)

SUMMARY:
The study objective is to establish feasibility of implementing a psychologically informed rehabilitation strategy while concurrently assessing its' effectiveness in Active duty service members (ADSM) with musculoskeletal disorders (MSD) seeking care in a US Navy shore-based healthcare setting. This intervention is intended to improve the management of chronic pain in order to optimize ADSM function.

The study team is proposing an observational prospective comparative cohort study. This study tests an implementation/strategy while observing/gathering information on the clinical intervention and related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ADSM (at baseline; separation from the military post-treatment will not be grounds for exclusion)
* Patients presenting to an NMCP or a branch clinic physical therapy department
* Patients who have only receive their evaluation appointment for their primary complaint
* Patients prescribing for a primary complaint of a MSD (the following ICD-10 codes will be included: M13, M14.8, M15-19, M21-25, M40-43, M46-48, M50-54, M60-71, M73, M75-77)

Exclusion Criteria:

* Patients not eligible to receive outpatient physical therapy
* Patients receiving fewer than four treatment sessions of physical therapy
* Patients who are pregnant
* Patients receiving physical therapy for acute post-surgical recovery
* Patients scheduled for or subject to a Physical Evaluation Board (PEB) at baseline
* Coast Guard

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: US active duty service members (ADSM) receiving physical therapy for musculoskeletal disorders at Naval Medical Center Portsmouth (NMCP) and its branch health clinics.
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Campello, PT, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to marco.campello@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-Training Arm (Control) | Post-Training Arm (Intervention)
Started | 219 | 208
Completed | 73 | 79
Not Completed | 146 | 129
Not completed — Withdrawal by Subject | 14 | 8
Not completed — Lost to Follow-up | 132 | 121

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Training Arm (Control) | Post-Training Arm (Intervention) | Total
Number analyzed (Participants) | 219 | 208 | 427
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (9) | 32 (8) | 32 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 85 | 173
  Male | 131 | 123 | 254
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 35 | 76
  Not Hispanic or Latino | 177 | 167 | 344
  Unknown or Not Reported | 1 | 6 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 9
  Asian | 11 | 11 | 22
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 67 | 70 | 137
  White | 122 | 120 | 242
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 12 | 0 | 12
Region of Enrollment [Number; unit: participants]
  United States | 219 | 208 | 427

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Disability Index (PDI) Score
Description: PDI consists of 7 categories of life activity. The participant is asked to circle the number on the scale that describes the level of disability on typically experiences. A score of 0 means no disability at all, and a score of 10 signifies that all of the activities in which one would normally be involved have been totally disrupted or prevented by pain. The total range of score is 0-70; the higher the score, the greater the person's disability due to pain.
Time Frame: Baseline, Follow-up 4 weeks
Population: Not all participants completed the follow-up questionnaire in full. Participants who did not complete the measure or only completed one measure but not others were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Change in PDI score
Arm/Group | Pre-Training Arm (Control) | Post-Training Arm (Intervention)
Number analyzed (Participants) | 71 | 70
Change in PDI score | 0 (11) | 33 (10)

2. Secondary Outcome: Change in Pain Catastrophizing Scale (PCS) Score
Description: PCS is a 13-item self-report measure designed to assess catastrophic thinking related to pain among adults with or without chronic pain. Each item is rated on a 5-point Likert scale, from 0 (not at all) to 4 (all the time). The total range of score is 0-52; a higher score indicates a higher level of catastrophizing. A total score >30 indicates clinically relevant level of catastrophizing.
Time Frame: Baseline, Follow-up 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in PCS score
Arm/Group | Pre-Training Arm (Control) | Post-Training Arm (Intervention)
Number analyzed (Participants) | 69 | 69
Change in PCS score | 0 (8) | 1 (7)

3. Secondary Outcome: Change in Hospital Anxiety and Depression Scale (HADS) Score
Description: HADS consists of two separate sub-sections: Anxiety and Depression. Each sub-section contains 7 items, where participants reply with responses that are closest to how he/she has been feeling in the past week with a score of 0-3. The total score range for both sub-sections is 0-21; a score of 0-7 indicates a "normal" range of anxiety, 8-10 = borderline abnormal, 11-21 = abnormal. The higher the score, the more abnormal the participant feels.
Time Frame: Baseline, Follow-up 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in HADS score
Arm/Group | Pre-Training Arm (Control) | Post-Training Arm (Intervention)
Number analyzed (Participants) | 69 | 69
Change in HADS score | -1 (5) | 0 (5)

4. Secondary Outcome: Change in Fear Avoidance Beliefs Questionnaire (FABQ) Score
Description: FABQ is a self-reported questionnaire consisting of 16 questions scaled from 0-6. FABQ assesses the fear-avoidance beliefs of patients with chronic low back pain The total range of score is 0-96; a higher score indicates fear avoidance behaviors. For the purposes of this study, "I have a claim for compensation for my pain" will be excluded due to no relevance to the study.
Time Frame: Baseline, Follow-up 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in FABQ score
Arm/Group | Pre-Training Arm (Control) | Post-Training Arm (Intervention)
Number analyzed (Participants) | 69 | 69
Change in FABQ score | -3 (11) | 1 (12)

5. Secondary Outcome: Change in Pain Self-Efficacy Questionnaire (PSEQ) Score
Description: PSEQ is a 10-item questionnaire developed to assess the confidence people with ongoing pain have in performing activities while in pain. The total range of score is 0-60; a higher score indicates greater levels of confidence in dealing with pain. High scores are strongly associated with clinically-significant functional levels.
Time Frame: Baseline, Follow-up 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in PSEQ score
Arm/Group | Pre-Training Arm (Control) | Post-Training Arm (Intervention)
Number analyzed (Participants) | 70 | 69
Change in PSEQ score | 0 (9) | 0 (13)

6. Secondary Outcome: MedRisk Instrument for Measuring Patient Satisfaction (MRPS) - Satisfaction With Process of Care Score
Description: Satisfaction with process of care is measured by the "process of care" subscale of the MRPS. There are 8 items in this subscale scored on a Likert scale of 1-5. The total score range is 8-40; the higher the score, the greater the satisfaction.
Time Frame: Follow-up 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pre-Training Arm (Control) | Post-Training Arm (Intervention)
Number analyzed (Participants) | 69 | 69
score on a scale | 32 (6) | 32 (6)

7. Secondary Outcome: Core Outcome Measures Index (COMI) - Satisfaction With the Outcome Score
Description: Satisfaction with the outcome is measured by a single item derived from COMI: "If you had to spend the rest of life with the symptoms you have right now, how would you feel about it?". The total range of score is 0-10; the higher the score, the worse one feels about the outcome.
Time Frame: Follow-up 4 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pre-Training Arm (Control) | Post-Training Arm (Intervention)
Number analyzed (Participants) | 68 | 68
score on a scale | 1 [1 to 2] | 2 [1 to 3]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Pre-Training Arm (Control) | Post-Training Arm (Intervention)
All-Cause Mortality (participants affected / at risk) | 0/219 | 0/208
Serious Adverse Events (participants affected / at risk) | 0/219 | 0/208
Other Adverse Events (participants affected / at risk) | 0/219 | 0/208

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT05132400/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT05132400/ICF_000.pdf